CLINICAL TRIAL: NCT00970099
Title: Mechanism of Exercise Training in Lean Insulin-Resistant Non-Diabetics
Brief Title: Mechanism of Insulin-Resistant in Lean Non-Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Ira Goldfine, UCSF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H6820-22194; 1R01DK059358-01A2 (NIH)
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Insulin Resistance; Insulin Sensitivity; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Active Comparator): 12 week exercise regimen
  Interventions: Behavioral: exercise
- non-exercise (Placebo Comparator): Normal lifestyle routine with no exercise for 12 weeks.
  Interventions: Behavioral: Non exercise

INTERVENTIONS:
Behavioral: exercise — Patients exercise under supervision on either a treadmill, Stair Master, or LifeCycle apparatus. Exercise frequency, duration, and intensity will be incrementally increased to minimize the risk of injury. During weeks 1-3, you will exercise for 30 minutes 3 days per week at 70- 80 % of your maximum heart rate (MHR); weeks 4-7 will consist of exercising for 40 minutes 4 days per week at 70-80% of your MHR; and weeks 7-12 will consist of exercising for 45 minutes 4 days per week at 80-85% MHR
  Arms: Exercise
Behavioral: Non exercise — subjects randomized to this group will not undergo exercise training for 12 weeks supervised by exercise specialist
  Arms: non-exercise

SUMMARY:
The study is designed to test the following primary hypothesis:

* Aerobic exercise training will improve insulin sensitivity in insulin resistant subjects through changes in the major cellular signaling pathways and and/or their regulators.

Accordingly, the proposed study is designed to accomplish the following specific aims:

* Quantitate how exercise training improves insulin sensitivity and decreases cardiovascular risk factors in a general population of lean, nondiabetic, insulin resistant subjects. Effects on known cardiovascular risk factors including blood pressure and serum lipoproteins will be evaluated. Change in regional adiposity will also be measured
* Determine the effects of a program of regular aerobic exercise on in the insulin receptor signaling pathway. Biopsies of vastus lateralis muscle from insulin resistant subjects will be obtained before and after a hyperinsulinemic glucose clamp. This procedure will take place in the untrained state and after exercise training. The investigators will measure changes in the insulin receptor and the activity of the major components of the intracellular insulin signaling pathway. The investigators will also look intracellular proteins that regulate this signaling pathway.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20-50
* No regular exercise for past 2 years

Exclusion Criteria:

* Diabetes, Cardiovascular disease, Pregnant or lactating females,BMI >27
* Medications that may interfere with carbohydrate metabolism - glucocorticoids, adrenergic agonists, ACE inhibitors, alpha blockers, diuretics, beta blockers, oral contraceptives, HMG CoA reductase inhibitors
* History of epilepsy, cancer, hepatitis, active infection, active Graves' disease, cystic fibrosis, sickle cell anemia, peripheral vascular disease, cerebrovascular disease, asthma
* Any medical condition that in the opinion of the investigator will interfere with safe completion of the trial
* Inability to give informed consent
* Prior participation in a clinical trial that could potentially alter insulin sensitivity: e.g., use of new insulin sensitizers
* HIV seropositive
* Anemia (Hgb < 12 g/dl)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2004-02; Primary Completion 2007-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity and insulin signaling | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ucsf Gcrc, San Francisco, California, United States